CLINICAL TRIAL: NCT03954405
Title: Multi-marker Approach for Risk Assessment in Pulmonary Arterial Hypertension (PAH)
Brief Title: Multi-marker Approach for Risk Assessment in PAH
Acronym: MARS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wuhan Asia Heart Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2018LMC-1
Record Dates: First submitted 2019-05-10; First posted 2019-05-17 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-01

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective registry including incident patients and prevalent patients which pretends to identify clinical characteristics, treatment trends in-hospital and ten years follow-up outcome through major adverse cardiovascular events (MACE) in a China population with well characterized PAH.

DETAILED DESCRIPTION:
baseline include: An echocardiogram to assess the size, shape, pumping action and the extent of any damage to the heart.

Lung function tests which include blowing measurements to assess gas volumes within the lungs as well as assessment of how the lungs exchange gases.

Right heart catheterisation (RHC) to diagnose PAH Optional Cardiac Magnetic Resonance tests. 6 minute walk distance (6MWD). To measure exercise capacity Electrocardiogram (ECG), a test that measures the electrical activity of the heart Blood tests

MACE include:

death heart/lung transplantation atrial septostomy hospitalization due to worsening of PAH start of new specific PAH treatment persistent decrease of >15% from baseline in 6MWD (or >30% compared with last study-related measurement) persistent worsening of World Health Organization (WHO) Functional Class (FC）

ELIGIBILITY:
Inclusion Criteria:

diagnosis of PAH (by RHC)

Exclusion Criteria:

Refusal to participate.

Ages: 1 Year to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with diagnosis of PAH from groups I
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
survival | 5 years
  To recruit a cohort of group 1 PAH cases. define the death as the primary outcome

SECONDARY OUTCOMES:
clinical worsening | 5 years
  one of the following: death, heart/lung transplantation, atrial septostomy, hospitalization due to worsening of PAH, start of new specific PAH treatment, persistent decrease of >15% from baseline in 6MWD (or >30% compared with last study-related measurement), persistent worsening of WHO FC

CONTACTS AND LOCATIONS:
Overall Officials: Qiu Qiu, Principal Investigator — Wuhan Asian Heart Hospital
Locations (1):
- Wuhan Asian Heart Hospital, Wuhan, China